CLINICAL TRIAL: NCT07262489
Title: Neo-adjuvant Adaptive Master Trial for Localized Cancers With Rapid Evaluation of Molecular & Immune Status for Stratified Immunotherapies in Oncology
Brief Title: Neo-adjuvant Immunotherapy Master Trial for Localized Cancers
Acronym: NEOREM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UC-IMM-2509; 2025-522127-95-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-24; First posted 2025-12-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Localized Cancer
Keywords: Neo-adjuvant immunotherapy; Localized cancers; Tumor biology

STUDY DESIGN:
Intervention Model Description: NEOREM includes a series of Phase 2 clinical trials that are not randomized. These trials are testing new immunotherapy strategies for localized solid malignancies that are eligible to receive neo-adjuvant therapy and have medical unmet needs related to disease-free survival, overall survival or quality of life. Each patient will undergo PORTRAIT immune profiling before starting neoadjuvant treatment, and again during treatment (at the time of surgery), using fresh blood and tumor tissue samples. This is done to closely study the biological features of the tumor. The progress of the disease and how well the treatment is working will be monitored through medical imaging and evaluated using RECIST v1.1 criteria-a standard method used to measure how tumors respond to treatment. After surgery, a standard adjuvant treatment (an additional therapy to help prevent the cancer from returning) may be recommended by the doctor. Patients will be followed for up to five years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm immunotherapy in Localized Cancers (Experimental): Each therapeutic sub-protocol will mention the description of the intervention(s) administered
  Interventions: Drug: Each therapeutic NEOREM sub-protocol will mention the description of intervention

INTERVENTIONS:
Drug: Each therapeutic NEOREM sub-protocol will mention the description of intervention — Each therapeutic NEOREM sub-protocol will mention the description of intervention

SUMMARY:
Most cancer treatments are developed without knowing whether the drug's targets are actually present in a patient's tumor or whether the patient is likely to benefit from the treatment. In addition, the immune environment surrounding the tumor changes significantly during the course of the disease, and the body's immune response to cancer tends to become less effective in later stages.

Currently, standard blood tests provide only basic information about a patient's immune, inflammatory, and metabolic systems. These tests do not offer a comprehensive picture of how each person's immune system is functioning. Similarly, traditional tests on tumor samples-which require frozen or preserved tissue and take a long time to process-are not fast enough to guide treatment decisions during clinical trials.

NEOREM is a "Master Protocol" which includes multiple therapeutic sub-protocols testing new immunotherapy strategies. (Immunotherapy is a type of cancer treatment that helps the immune system fight cancer.) Neoadjuvant immunotherapies are treatments given before surgery. Their goals are to shrink the tumor to make it easier to remove, strengthen the immune system's ability to fight cancer, increase the chances of long-term recovery, and reduce the risk of the cancer returning.

This master protocol focuses on cancers that are still localized (have not spread) and aims to personalize treatments based on each patient's individual immuno-biological profile. As a part of this master protocol, a rapid analysis called PORTRAIT-which stands for "Profile in Onco-Immunology for a Rapid Treatment Research Adapted to Immunity and Tumor"-will be performed using fresh blood and tumor samples from each patient. This profiling uses highly sensitive and specific techniques to accurately detect biological markers that can predict how well someone will respond to immunotherapy before surgery.

NEOREM's overall goal is to test new treatment strategies and new methods of selecting patients (using the PORTRAIT immune profiling) to improve the effectiveness of current standard treatments for certain types of cancer while also reducing their side effects.

DETAILED DESCRIPTION:
Most cancer treatments are developed without knowing whether the drug targets are present in the tumors of patients enrolled in clinical trials or whether the patients have the tumor biology needed to benefit from such treatments. Tumor biology evolves as cancer progresses, resulting in weaker immune responses in advanced stages.

Traditional tumor analyses rely on formalin-fixed, paraffin-embedded (FFPE) or frozen materials for techniques such as immunohistochemistry (IHC) or DNA/RNA sequencing, which require long turnaround times. Routine blood tests provide only basic information about a patient's immune, inflammatory, and metabolic status, without offering detailed insight into the immune system. Research shows that analyzing fresh tumor and blood samples better predicts immunotherapy responses, supports patient monitoring, and helps identify biological subgroups that may benefit from new treatments.

The PORTRAIT method (Profile in Onco-Immunology for a Rapid Treatment Research Adapted to Immunity and Tumor) reduces turnaround time for biological analyses within NEOREM. It allows patients and oncologists to access relevant tumor and blood information at the molecular and cellular levels, identify appropriate treatment options, and assess treatment effects on the disease. PORTRAIT uses multicolor flow cytometry on fresh mononuclear cells from patient blood and tumor biopsies to screen for specific biomarkers. Plasma and tumor secretome are analyzed for cytokines, chemokines, and soluble factors to provide a comprehensive immune and tumor profile. This approach helps determine which patients are eligible for specific treatments within the sub-protocols.

NEOREM is part of the REMISSION program, which includes a Master Protocol linked to therapeutic sub-protocols. The Master Protocol provides a unified framework to test multiple study drugs efficiently, streamline operations, optimize resources, and accelerate patient access to treatments. Its flexible design allows sub-protocols to be added or closed quickly without affecting ongoing studies, while adaptive analytics integrate evidence across studies to maximize knowledge and leverage historical data. Standardized processes, centralized data infrastructure, and consistent recruitment centers further improve safety, data quality, and operational efficiency.

The goal of the NEOREM protocol is to improve cancer care by accelerating the development of neoadjuvant immunotherapy strategies. These therapies leverage pre-existing tumor-infiltrating lymphocytes (TILs) and draining lymph nodes before surgery to strengthen the antitumor immune response. Neoadjuvant therapy may downstage localized tumors, simplify surgery, achieve complete responses, sometimes eliminate the need for major procedures, improve quality of life, and reduce the risk of recurrence.

PORTRAIT immunoprofiling from fresh blood and tumor samples provides a rapid and detailed description of each patient's immune profile. This enables a deeper understanding of disease biology and allows patients to be quickly stratified into the most appropriate therapeutic sub-protocol, supporting truly personalized cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 12 years with at least 40kg body weight or otherwise as per specified in sub-protocol.
2. Prior to the inclusion in the NEOREM master protocol, patients must have signed a written informed consent to baseline PORTRAIT profiling.

   Note:
   * When the patient is physically unable to give his/her written consent, a trusted person of his/her choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent.
   * For patients aged between > 12 and < 18, specific consent from legal tutors should be obtained on top of the minor consent and prior procedures.
3. Localized solid malignancy that is eligible to receive neo-adjuvant therapy and has medical unmet needs related to disease-free survival, overall survival or quality of life.

   Note: Specific sub-protocols could enroll patients with inoperable tumors with the aim of downstaging them to become operable.
4. Having a measurable disease (i.e. at least one measurable lesion according to RECIST v1.1 for solid tumors.
5. Eastern cooperative oncology group (ECOG) performance status between 0 and 2.
6. Patients amenable to undergo blood draw and tumor biopsy procedures.
7. Adequate organ function as defined by the following criteria:

   * Total bilirubin ≤1.5 ULN, or ≤3.0 ULN in participants with Hepato-Cellular Carcinoma (HCC) or known Gilbert's syndrome if the increase is predominantly due to unconjugated bilirubin.
   * ALT ≤ 3 x ULN; if liver metastases ALT ≤ 5 x ULN
   * Absolute Neutrophils count (ANC) ≥ 1000 cells/mm³ in the absence of G-CSF or GM-CSF within ≤2 weeks before the first dose of trial treatment.
   * Platelets ≥100 000 cells/mm³
   * Hemoglobin ≥ 9.0 g/dL
   * Albumin ≥ 30 g/L
   * Calculated creatinine clearance ≥50 mL/min/1.73 m2
8. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment.
9. Both sexually active WOCBP and male (and their WOCBP partners) patients must agree to use two methods of effective contraception, one of them being a physical barrier method, or to abstain from sexual activity during the study and for the period indicated in specific sub-protocol after the last study drug administration.
10. Patient affiliated to the French social security regimen.
11. Patients with mental and legal ability to fully consent for undergoing the exploratory procedures (blood draws and biopsies) prior and upon treatment (at baseline PORTRAIT and once on-treatment PORTRAIT).
12. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. Cancer patients with advanced stages and/or distant metastasis (unless curable oligometastatic disease). Some sub-protocols could enroll patients with loco-regional (N+) stages amenable to curative intention strategies.
2. Any life-threatening allergy to one of the experimental products tested in the sub-protocol where the patient is eligible. In case of allergy to contrast media, patient monitoring should be performed with alternate methods (both CT-scan or MRI).
3. History of life threatening autoimmune/immune mediated inflammatory disease, including but not limited to severe colitis, pneumonitis, Guillain-Barré syndrome, anti-phospholipid syndromes and myocarditis. Patients with a history of auto-immune endocrinopathy (hypo/hyper thyroiditis, type 1 diabetes mellitus, …) and who are stable on hormone replacement therapy are eligible for the study. Patients with a history of vitiligo, alopecia areata, cutaneous psoriasis and grade 1-2 Sjogren syndrome are eligible.
4. Treatment with systemic long-term immunosuppressive medications unless otherwise specified in the specific therapeutic sub-protocols. Those immunosuppressive drugs must have been stopped at least 4 weeks prior to enrolment. Hormone replacement therapy with physiological doses of hydrocortisone is acceptable.
5. Chemotherapy, hormonotherapy, radiotherapy or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks or 5 half-life times (whatever the shortest) prior to treatment with the trial drugs.
6. Administration of a live, attenuated vaccine within 4 weeks prior to enrolment.
7. Radiotherapy to the chosen RECIST target lesion(s) (unless a progression after radiotherapy has been documented).
8. Persistence of a clinically relevant treatment-related toxicity from previous chemotherapy, targeted therapy and/or local treatments which could hamper the safety or efficacy assessment of the therapy tested (for previous disease).
9. Patients with evolving tumors next to cavitary or major blood vessels at high risk of massive bleeding and/or perforation.
10. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial.
11. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned major surgery during the on-treatment study period.
12. History of clinically significant hemorrhagic or thromboembolic event in the past 3 months.
13. History of significant cardiovascular diseases (i.e. supraventricular tachycardia, uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion).
14. Ongoing uncontrolled endocrinopathy. Ancient endocrinopathy currently stable with substitutive therapy should not be excluded from the trial.
15. Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix. A history of more than 3 years of local prostate cancer treated by surgery and without PSA elevation since surgery, or local breast carcinoma treated by surgery without relapse or resected non-muscle invasive bladder cancers are eligible.
16. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy. A wash out of more than 3 weeks is required after last systemic antibiotics to allow reconstitution of the microbiome. Patients infected by HIV but having efficient anti-retroviral therapy and CD4+ T-cell counts >500/mm³ are eligible. Patients with a history of HBV or HCV that are cured and have eligible liver function criteria are also eligible.
17. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug in case an oral drug is tested in the sub-protocol for which the patient is screened.
18. Pregnancy or breastfeeding.
19. Intake of Ganoderma Lucidum mushroom (also called "Reishi") and/or herbal remedies and/or traditional medicines within the past weeks prior to start of trial treatment or concomitantly with the trial because of their potential to increase treatment related adverse events.
20. Any psychological, familial, sociological, geographical factors, lifestyle, behavior, clinical or biological parameters or elements in the past medical history of the patients that, according to the investigator, could preclude the ability of the trial to directly reach its objectives, or indirectly via treatment observance or study follow up. Patients with active alcoholism and/or drug abuse are excluded.
21. Person deprived of its liberty or under protective custody or guardianship.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
The main objective is to evaluate efficacy of novel treatment strategies to increase the patient population therapeutic index in histology-based or tumor-agnostic/biomarker-driven oncology indications | Through all the NEOREM subprotocols completion and no new subprotocol is designed, an average of 7 years
  In the context of NEOREM, increasing the therapeutic index means enhancing the effectiveness of a treatment strategy-measured through efficacy endpoints - as complete pathological response,pCR, defined as the complete absence of viable tumor cells or major pathological response i.e. less than 10% viable tumor cells in the surgical specimen - within patient groups most likely to benefit, while reducing toxicity risks in those unlikely to respond.
The main objective is to evaluate safety of novel treatment strategies to increase the patient population therapeutic index in histology-based or tumor-agnostic/biomarker-driven oncology indications | Through all the NEOREM subprotocols completion and no new subprotocol is designed, an average of 7 years
  Safety measurements will include the percentage of patients whose surgery was delayed beyond the planned timeline, due to treatment-related adverse events.
The main objective is to evaluate patient selection criteria to increase the patient population therapeutic index in histology-based or tumor-agnostic/biomarker-driven oncology indications | Through all the NEOREM subprotocols completion and no new subprotocol is designed, an average of 7 years
  The sub-protocols may be designed as exploratory or confirmatory trials to validate immune biomarkers for patient selection using PORTRAIT immunoprofiling. PORTRAIT profiling can be generated on from fresh whole blood and fresh tumor biopsies in order to allow for a rapid, sensitive and specific description of each patient's immuno-biological profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France